CLINICAL TRIAL: NCT04917796
Title: A Randomized Phase III Clinical Trial of Acupuncture for Chemotherapy-induced Peripheral Neuropathy Treatment (ACT)
Brief Title: The Effect of Electroacupuncture on Nerve Pain Caused by Chemotherapy (Chemotherapy-Induced Peripheral Neuropathy)
Acronym: ACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Ting Bao, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-510
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Nerve Pain; Neuropathy; Neuropathy, Painful; Pain; CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Chemotherapy-induced Peripheral Neuropathy; CIPN; Electroacupuncture; Cancer survivor; Acupuncture; Memorial Sloan Kettering Cancer Center; Neuropathy; Dana-Farber Cancer Institute; Neuropathic Pain; Pain Management
MeSH Terms: conditions — Neuralgia; Neuropathy, Painful; Pain; Agnosia | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization will occur before the baseline assessments are administered. Each site will randomize its own patients through RedCap. Once the patient is randomized, the site acupuncture team will be notified via RedCap alert in order to provide the appropriate treatment. Patients and non-acupuncturist members of the study team will be blinded to which acupuncture group the patient was assigned. The acupuncturists and one clinical research coordinator will be the only ones unblinded. The clinical research coordinator will be unblinded in order to assist acupuncturists to confirm randomization. This clinical research coordinator will not be the primary research coordinator in the study and will not have direct contact with the patient. The rest of the study coinvestigators and staff will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture Arm (Experimental): The study participants will include 250 cancer survivors who have completed neurotoxic agent containing chemotherapy at least three months prior and have persistent moderate to severe Chemotherapy-Induced Peripheral Neuropathy/CIPN pain randomized to one of two study arms.
  Interventions: Other: Electroacupuncture
- Sham Acupuncture Arm (Placebo Comparator): The study participants will include 250 cancer survivors who have completed neurotoxic agent containing chemotherapy at least three months prior and have persistent moderate to severe Chemotherapy-Induced Peripheral Neuropathy/CIPN pain randomized to one of two study arms.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Electroacupuncture — Real and sham acupuncture will be delivered by experienced licensed acupuncturists. The intervention includes 10 treatments of acupuncture over 8 weeks (i.e., twice per week for two weeks, then one treatment per week for six weeks).
  Other Names: EA
  Arms: Electroacupuncture Arm
Other: Sham Acupuncture — Real and sham acupuncture will be delivered by experienced licensed acupuncturists. The intervention includes 10 treatments of acupuncture over 8 weeks (i.e., twice per week for two weeks, then one treatment per week for six weeks).
  Arms: Sham Acupuncture Arm

SUMMARY:
This study is a randomized controlled trial of electroacupuncture (referred to as EA) versus sham acupuncture (referred to as EA) as effective treatments for Chemotherapy-Induced Peripheral Neuropathy (CIPN) pain in cancer survivors.

DETAILED DESCRIPTION:
During the study, patients will be randomized to one of the two possible acupuncture treatment groups and receive 10 treatments over the course of 8 weeks and then enter a follow-up period. Acupuncture is a medical technique that involves insertion of very thin needles into specific areas on the body with the goal of promoting health and well-being. EA involves adding a very small amount of electricity through the acupuncture needles (electrical stimulation). Researchers have found that EA can increase the effects of regular acupuncture, and it is particularly helpful for treating different kinds of pain. The purpose of this study is to learn if EA can improve CIPN pain in cancer survivors, and if it is effective against other CIPN-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient men and women aged ≥18 years
* Free of oncologic disease by clinical examination and history
* Completed neurotoxic chemotherapy such as platinum agents, taxanes, vinca alkaloids, and bortezomib at least three months prior to enrollment
* Diagnosis of CIPN based on symptom history, loss of deep tendon reflexes, or the presence of symmetrical stocking-glove pain, numbness, or paresthesia
* Grade ≥1 sensory pain based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* Self-reported moderate to severe CIPN pain, as defined by a score of 4 or greater on the BPI-SF average pain item over the past week
* On a stable regimen (no change in the past three months) if taking anti-neuropathy or other pain medications
* Willing to adhere to requirement that no new pain medication be taken throughout the first 12 weeks of the study period
* Willing to adhere to all study-related procedures, including randomization to one of the two possible acupuncture treatments

Exclusion Criteria:

* Patients with a pacemaker or other electronically charged medical device
* Use of acupuncture for symptom management within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Difference of pain severity from baseline to 4 weeks after baseline. | 4 weeks
  The primary outcome will be the patient's rating of his/her average pain in the past 24 hours. All participants will fill out the Brief Pain Inventory-Short Form (BPI-SF)
Difference of pain severity from baseline to 8 weeks after baseline. | 8 weeks
  The primary outcome will be the patient's rating of his/her average pain in the past 24 hours. All participants will fill out the Brief Pain Inventory-Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Ting Bao, MD at ting_bao@dfci.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- See also: Dana-Farber Cancer Institute — https://www.dana-farber.org/
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org